CLINICAL TRIAL: NCT06169579
Title: A Single-arm, Non-randomized, Open-label, Dose-escalation and Dose-expansion, Multicenter Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profiles, as Well as Preliminary Efficacy, of ND-003 in Chinese Patients With Advanced Solid Tumors.
Brief Title: An Open-label, Phase 1 Study to Determine the Maximum Tolerated Dose of ND-003 in Patients With Advanced Solid Cancers
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen NewDEL Biotech, Co., Ltd (Industry)
Collaborators: Shenzhen Innovation Center for Small Molecule Drug Discovery Co., Ltd. (Unknown); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ND-003-I
Record Dates: First submitted 2023-11-23; First posted 2023-12-13 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- ND-003 tablets_Dose 1 (Experimental): Adult patients with solid tumors receiving 40 mg of ND-003 tablets once daily (dose escalation cohort).
  Interventions: Drug: ND-003 tablets
- ND-003 tablets_Dose 2 (Experimental): Adult patients with solid tumors receiving 80 mg of ND-003 tablets once daily (dose escalation cohort).
  Interventions: Drug: ND-003 tablets
- ND-003 tablets_Dose 3 (Experimental): Adult patients with solid tumors receiving 160 mg of ND-003 tablets once daily (dose escalation cohort).
  Interventions: Drug: ND-003 tablets
- ND-003 tablets_Dose 4 (Experimental): Adult patients with solid tumors receiving 300 mg of ND-003 tablets once daily (dose escalation cohort).
  Interventions: Drug: ND-003 tablets
- ND-003 tablets_Dose 5 (Experimental): Adult patients with solid tumors receiving 500 mg of ND-003 tablets once daily (dose escalation cohort).
  Interventions: Drug: ND-003 tablets
- ND-003 tablets_Dose 6 (Experimental): Adult patients with solid tumors receiving 800 mg of ND-003 tablets once daily (dose escalation cohort).
  Interventions: Drug: ND-003 tablets
- ND-003 tablets_Expansion 1 (Experimental): Adults patients with solid tumors harboring NTRK or RET Fusion or Mutation (dose expansion cohort).
  Patients receive either the recommended or maximum tolerated dose of ND-003 tablets as determined in the dose escalation part, one to two dose cohorts are set.
  Interventions: Drug: ND-003 tablets
- ND-003 tablets_Expansion 2 (Experimental): Adults patients with solid tumors harboring NTRK or RET Fusion or Mutation (dose expansion cohort).
  Patients receive either the recommended or maximum tolerated dose of ND-003 tablets as determined in the dose escalation part, one to two dose cohorts are set.
  Interventions: Drug: ND-003 tablets

INTERVENTIONS:
Drug: ND-003 tablets — ND-003 tablets will be administered orally and observe 4 days, and followed by over continuous 28-days cycles.
  Other Names: ND003 tablets
  Arms: ND-003 tablets_Dose 1
Drug: ND-003 tablets — ND-003 tablets will be administered orally and observe 4 days, and followed by over continuous 28-days cycles.
  Other Names: ND003 tablets
  Arms: ND-003 tablets_Dose 2
Drug: ND-003 tablets — ND-003 tablets will be administered orally and observe 4 days, and followed by over continuous 28-days cycles.
  Other Names: ND003 tablets
  Arms: ND-003 tablets_Dose 3
Drug: ND-003 tablets — ND-003 tablets will be administered orally and observe 4 days, and followed by over continuous 28-days cycles.
  Other Names: ND003 tablets
  Arms: ND-003 tablets_Dose 4
Drug: ND-003 tablets — ND-003 tablets will be administered orally and observe 4 days, and followed by over continuous 28-days cycles.
  Other Names: ND003 tablets
  Arms: ND-003 tablets_Dose 5
Drug: ND-003 tablets — ND-003 tablets will be administered orally and observe 4 days, and followed by over continuous 28-days cycles.
  Other Names: ND003 tablets
  Arms: ND-003 tablets_Dose 6
Drug: ND-003 tablets — ND-003 tablets will be administered orally over continuous 28-days cycles.
  Other Names: ND003 tablets
  Arms: ND-003 tablets_Expansion 1
Drug: ND-003 tablets — ND-003 tablets will be administered orally over continuous 28-days cycles.
  Other Names: ND003 tablets
  Arms: ND-003 tablets_Expansion 2

SUMMARY:
This study is done to test the safety and preliminary efficacy of drug ND-003 tablets in patients with solid tumors. ND-003 is a highly potent and selective small molecular inhibitor of NTRK (neurotrophic receptor tyrosine kinase) and RET (rearranged during transfection). The study also investigates how the drug is absorbed and processed in the human body.

DETAILED DESCRIPTION:
The trial will be conducted in 2 parts: an initial dose escalation phase of drug ND-003 tablets in patients with solid tumors will be followed by an expansion phase in subjects with solid tumors harboring NTRK or RET Fusion or Mutation.

The objectives of the study are to determine the safety, tolerability, pharmacokinetic and pharmacodynamics profiles, as well as preliminary efficacy of orally administered ND-003 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with advanced malignant solid tumors confirmed by histology or cytology.
2. Subjects have previously received standard treatment with failure (including disease progression or toxicity intolerance), or have no available standard treatment plans, or have contraindications to standard treatment.
3. In the dose escalation phase, NTRK or RET gene fusion status is not an eligibility criterion, but subjects harboring NTRK or RET fusion or mutation will be prioritized. However, in the dose expansion phase, subjects must have confirmed NTRK or RET gene fusion/mutation (histologic or cytological genetic testing results are acceptable) .
4. Patients have at least one evaluable lesion according to RECIST version 1.1 evaluation criteria ( Revised RECIST Guidelines (version 1.1) );
5. Subjects must be 18 years or older (no limitation by sex or maximum age) on the day of signing informed consent .
6. Have an Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 2.
7. Have a projected life expectancy of at least 12 weeks .
8. Have adequate organ and bone marrow function to meet laboratory examination standards.
9. Fertile male subjects and childbearing potential female subjects agree to use highly effective contraception from the time of signing informed consent until 6 months after the final dose of investigational product. Childbearing potential female subjects include premenopausal women and women within 2 years after menopause; Pregnancy testing results for childbearing potential female subjects within ≤ 7 days before the first administration must be negative.
10. Capable of understanding the written informed consent document; willingly provides valid, signed written informed consent; willing and able to comply with the schedule, requirements and restrictions of the study.

Exclusion criteria:

1. Known hypersensitivity to ND-003 or any of its constituents.
2. Previous exposure to ND-003.
3. Subjects participated or are currently participating in clinical trials of other drugs or medical devices within 4 weeks prior to the first administration.
4. Subjects underwent major surgery within 4 weeks before the first administration or had a surgical plan during the study period.
5. Received systemic anti-tumor drug therapy such as chemotherapy, macromolecular targeted therapy, endocrine therapy within 3 weeks before the first administration (subjects have previously used nitrosourea or mitomycin C with a washout period of at least 6 weeks; subjects have previously used oral fluorouracil drugs or small molecule targeted drugs with a washout period of at least 2 weeks or 5 half-lives, whichever is the longer.) or radiation therapy, or immunotherapy within 4 weeks before administration.
6. Use traditional Chinese patent medicines with anti-tumor effect within 2 weeks before the first administration.
7. Receipt of live vaccine within 4 weeks prior to study drug administration or plan to receive them during the study period, including but not limited to: measles, mumps, rubella, chickenpox, yellow fever, rabies, Bacillus calmette-guerin (BCG) and typhoid vaccines.
8. Subjects who used known concomitant drugs that can prolong the QT interval and/or CYP2C8, CYP3A strong inhibitors and/or inducers within 7 days before the first administration, as well as those who need to continue using the aforementioned drugs during the study period.
9. Subjects who have suffered from another type of malignant tumor within the past 5 years, excluding those who have received curative treatment for cervical cancer in situ, non melanoma skin cancer, localized prostate cancer, ductal cancer in situ, and other extremely low-risk malignant tumors.
10. Loss or donation of blood > 500 mL (within 3 months before the first administration).
11. Donation of bone marrow or peripheral stem cells (within 3 months before the first administration).
12. Uncontrolled or symptomatic central nervous system (CNS) metastasis including symptomatic brain metastasis or meningeal metastasis or spinal cord compression; but the following patients are allowed to be included: a. subjects with treated brain metastasis (such as surgery or radiation therapy), there was no progress in imaging and/or no neurological symptoms or signs appeared after treatment at least 4 weeks before the first administration, there was no evidence of new brain metastasis or increased metastasis, and systemic hormone therapy (dosage>10 mg/day of prednisone or other effective hormones) was stopped at least 4 weeks before the first administration; b. Untreated and asymptomatic subjects with brain metastases do not require corticosteroids, and the length of brain metastases are ≤ 1.5 cm.
13. Suffering from uncontrollable diseases, including but not limited to:

1）Existence of persistent or active infections (including bacteria, fungi, viruses, etc.) that require antibiotic, antifungal, or antiviral treatment; 2）Acute coronary syndrome, congestive heart failure (New York Heart Association Cardiac Function Classification ≥ Level II), left ventricular ejection fraction (LVEF)<50%, cerebrovascular accident, transient ischemic attack, stroke, deep vein thrombosis, pulmonary embolism, aneurysm, arterial dissection, or other level 3 or above cardiovascular and cerebrovascular events occurred within 6 months before the first administration; 3）Investigator considers that arrhythmias (such as bradycardia) with clinical significant or conduction abnormalities, congenital long QT interval syndrome or Fridericia's corrected QTc (corrected QT interval) are unmeasurable or QTcF>450 msec; 4）Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) or hypotension (systolic blood pressure less than 80 mmHg and/or diastolic blood pressure less than 50 mmHg); 5）Uncontrolled hyperglycemia; 6）Active peptic ulcer disease or gastritis, active hemorrhagic disease; 7）Mental illness/social conditions that affect patients' compliance with clinical trials and their ability to sign written informed consent forms.

14.Have family history of long QT syndrome or unexplained sudden death in first degree relatives under the age of 40.

15.Unable to swallow medication orally, have gastrointestinal abnormalities with clinical significant (such as after gastrointestinal resection, gastrointestinal anastomosis, chronic diarrhea, and intestinal obstruction), or have significant impact on gastrointestinal absorption as determined by the investigator 16.Individuals with difficulty in venous blood collection (such as fainting or fainting history due to syringe) 17.History of drug or alcohol abuse . 18.Human immunodeficiency virus (HIV) antibodies positive or active syphilis or active pulmonary tuberculosis (determined by the investigator based on the tuberculin test or γ- Interferon release test [T-SPOT test] results, imaging examination results and comprehensive judgment of clinical symptoms) or hepatitis C virus antibody positive and hepatitis C virus (HCV) RNA positive, or active hepatitis B patients (hepatitis B surface antigen positive and HBV (Hepatitis B virus honeybee venom) DNA ≥ the upper limit of normal value).

19.Failure to recover from any AE related to previous surgical procedures and previous cancer treatment (CTCAE 5.0 rating to ≤ 1), except for the following situations: a. hair loss; b. Level 1 toxicity without clinical significance, such as lymphopenia.

20.Pregnant or lactating women, or planning to conceive during the study period.

21.Investigator considers that the subjects may have other situations that may affect compliance or may not be suitable to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | 4 days after single oral administration and the first cycle of multiple administration (28 days)
  DLT is defined as adverse events (graded according to NCI CTCAE ver5.0) assessed by the investigator to be definitely/probably/possibly related to the investigational product
Maximum tolerated dose (MTD) | 4 days after single oral administration and the first cycle of multiple administration (28 days)
  MTD is defined as the highest dose level at which fewer than 1 of 6 subjects experienced DLT.
Adverse Events (AE) assessed by CTCAE ver5.0. | through study completion, an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE ver5.0.

SECONDARY OUTCOMES:
maximum concentration (Cmax) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours after at a singe dose administration of ND-003
  The drug maximum concentration reaches when the absorption rate is equal to the elimination rate at a single dose.
Time to maximum concentration (Tmax) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours after at a singe dose administration of ND-003
  Time required to reach peak drug concentration after a single administration.
Elimination Half-life (t1/2) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours after a single dose administration.
  Elimination Half-life (t1/2) refers to the time required to eliminate 50% of the drug from the body.
Clearance (CL/F) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours after a single dose administration.
  Clearance (CL) describes how the body effectively eliminate drugs from the systemic circulation, typically defined as the volume of drug-containing plasma eliminated from the body per unit time.
AUC from time 0 to last time of quantifiable concentration (AUC0-t) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours after a single dose administration.
  Area under the plasma concentration-time curve from the initial administration to the last measurable concentration point
Objective response rate (ORR) | Baseline through up to 6 cycles or until disease progression (each cycle is 28 days)
  ORR is defined as confirmed complete response (CR) or partial response (PR) based on RECIST (version 1.1) .
Progression-free survival (PFS) | Baseline through up to 6 cycles or until disease progression (each cycle is 28 days)
  PFS is defined as the time from randomization until objective tumor progression or death, whichever occurs first.
Overall survival (OS) | Baseline through up to 6 cycles or until disease progression (each cycle is 28 days)
  Overall survival is defined as the time from randomization until death from any cause and is measured in the intent-to-treat population.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PhD, Principal Investigator — Sun Yat-sen University
Locations (21):
- China (21):
  - the First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - the first hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen University cancer center, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Zhanjiang Central Hospital, Guangdong Medical University, Zhanjiang, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - the Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Tongji Hospital Tongji Medical College of HUST, Wu’an, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Cancer Hospital & Institute, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - The Second People's Hospital of Neijiang, Neijiang, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang